CLINICAL TRIAL: NCT03948737
Title: The Effect of Alpha-tocopherol in Hemolysis and Oxidative Stress Marker on the Red Cell
Brief Title: The Effect of Alpha-tocopherol in Hemolysis and Oxidative Stress Marker on the Red Cell Membrane Beta-thalassemia Major
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nora Sovira, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSovira
Record Dates: First submitted 2019-05-07; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Beta Thalassemia Major Anemia; Hemolysis; Oxidative Stress
Keywords: Haptoglobin; Hemopexin; Hemolysis; Malondialdehyde; Glutathione; Oxidative stress; Alpha-Tocopherol
MeSH Terms: conditions — Hemolysis | interventions — alpha-Tocopherol

STUDY DESIGN:
Intervention Model Description: Beta thalassemia major children
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double masking. No any information about treatment or placebo in participant, investigator, care provider and outcome assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha-Tocopgerol (Active Comparator): Alpha-Tocopherol supplementation will be given orally for 4 weeks with doses adjusted by age.
  5-8 years old: 200 mg daily, 9-13 years old: 400 mg daily and 14-18 years old 600 mg daily.
  Interventions: Drug: Alpha-Tocopherol; Drug: Placebo oral tablet
- Control (Placebo Comparator): Placebo is the drug with the same shape and color as the alpha-tocopherol supplementation.
  Interventions: Drug: Alpha-Tocopherol; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Alpha-Tocopherol — all of the subjects in the alpha-tocopherol group received alpha-tocopherol orally, doses adjusted by age for 4 weeks of treatment.
  Other Names: Santa E
Drug: Placebo oral tablet
  Other Names: Alpha-tocopherol placebo

SUMMARY:
The accumulation of unpaired α-globin chains in β-thalassemia major patients may clinically create ineffective erythropoiesis, hemolysis, and chronic anemia. Multiple blood transfusions and iron overload cause cellular oxidative damage. However, α-tocopherol, an antioxidant, has been known as a potent scavenger of lipid radicals in the red cell membrane of β-thalassemia major patient. By this randomized controlled trial, the investigators would like to evaluate the effects of α-tocopherol in hemolysis and oxidative stress on the red cell membrane of β-thalassemia major.

DETAILED DESCRIPTION:
Background: The accumulation of unpaired α-globin chains in β-thalassemia major patients may clinically create ineffective erythropoiesis, hemolysis, and chronic anemia. Multiple blood transfusions and iron overload cause cellular oxidative damage. However, α-tocopherol, an antioxidant, has been known as a potent scavenger of lipid radicals in the red cell membrane of β-thalassemia major patients.

Purpose: To evaluate the effects of α-tocopherol in hemolysis and oxidative stress on the red cell membrane of β-thalassemia major.

Methods: In this randomized controlled trial, the investigators allocated subjects in the placebo and α-tocopherol groups. Doses of α-tocopherol were based on the recommendation of Institute of Medicine: 4-8 years old 200 mg/day; 9-13 years old 400 mg/day; 14-18 years old 600 mg/day. Hemolysis, oxidative stress, and antioxidant variables were evaluated before and after 4 weeks of consuming either α-tocopherol or placebo, performed prior to blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* received frequent transfusions,
* iron chelation
* aged 5 - 18-year-olds
* with no other hematologic disorders
* does not consume any other antioxidants or herbal supplements

Exclusion Criteria:

* the acute or chronic infection including hepatitis B or hepatitis C,
* splenectomy
* liver failure
* abnormality level of lipid test

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
The effects of α-tocopherol in hemolysis marker on the red cell membrane of β-thalassemia major | 4 weeks
  The plasma haptoglobin and hemolysis as hemolysis marker on alpha-tocopherol treatment were assessed by ELISA using Haptoglobin and Hemopexin kit for human

SECONDARY OUTCOMES:
The effects of α-tocopherol in oxidative stress marker on the red cell membrane of β-thalassemia major | 4 weeks
  The malondialdehyde plasma level as oxidative stress marker on alpha-tocopherol treatment was assessed by Spectrophotometry using TBARS method.
The effects of α-tocopherol in endogenous antioxidant on the red cell membrane of β-thalassemia major | 4 weeks
  The Glutathione as endogenous antioxidant marker on alpha-tocopherol treatment was assessed by ELISA method by using GT40 for Glutathione kit

CONTACTS AND LOCATIONS:
Overall Officials: Pustika Amalia, Consultant, Principal Investigator — Hematology Oncologist Head Division of Child Health of Universitas Indonesia
Locations (1):
- Thalassemia Centre Kiara RSUP Dr.CiptoMangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fibach E, Rachmilewitz EA. Pathophysiology and treatment of patients with beta-thalassemia - an update. F1000Res. 2017 Dec 20;6:2156. doi: 10.12688/f1000research.12688.1. eCollection 2017. PMID 29333256
- [Result] Voskou S, Aslan M, Fanis P, Phylactides M, Kleanthous M. Oxidative stress in beta-thalassaemia and sickle cell disease. Redox Biol. 2015 Dec;6:226-239. doi: 10.1016/j.redox.2015.07.018. Epub 2015 Aug 1. PMID 26285072
- [Result] Smith A, McCulloh RJ. Hemopexin and haptoglobin: allies against heme toxicity from hemoglobin not contenders. Front Physiol. 2015 Jun 30;6:187. doi: 10.3389/fphys.2015.00187. eCollection 2015. PMID 26175690
- [Result] Schaer CA, Deuel JW, Bittermann AG, Rubio IG, Schoedon G, Spahn DR, Wepf RA, Vallelian F, Schaer DJ. Mechanisms of haptoglobin protection against hemoglobin peroxidation triggered endothelial damage. Cell Death Differ. 2013 Nov;20(11):1569-79. doi: 10.1038/cdd.2013.113. Epub 2013 Aug 30. PMID 23995229
- [Result] Kormoczi GF, Saemann MD, Buchta C, Peck-Radosavljevic M, Mayr WR, Schwartz DW, Dunkler D, Spitzauer S, Panzer S. Influence of clinical factors on the haemolysis marker haptoglobin. Eur J Clin Invest. 2006 Mar;36(3):202-9. doi: 10.1111/j.1365-2362.2006.01617.x. PMID 16506966
- [Result] Schaer DJ, Vinchi F, Ingoglia G, Tolosano E, Buehler PW. Haptoglobin, hemopexin, and related defense pathways-basic science, clinical perspectives, and drug development. Front Physiol. 2014 Oct 28;5:415. doi: 10.3389/fphys.2014.00415. eCollection 2014. PMID 25389409
- [Result] Chow J, Phelan L, Bain BJ. Evaluation of single-tube osmotic fragility as a screening test for thalassemia. Am J Hematol. 2005 Jul;79(3):198-201. doi: 10.1002/ajh.20387. PMID 15981230
- [Result] Ghone RA, Kumbar KM, Suryakar AN, Katkam RV, Joshi NG. Oxidative stress and disturbance in antioxidant balance in beta thalassemia major. Indian J Clin Biochem. 2008 Oct;23(4):337-40. doi: 10.1007/s12291-008-0074-7. Epub 2008 Dec 20. PMID 23105782
- See also: Drug information of alpha-Tocopherol — https://druginfo.nlm.nih.gov/drugportal/name/alpha-Tocopherol+succinate

DOCUMENTS (1):
  • Study Protocol (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03948737/Prot_000.pdf